CLINICAL TRIAL: NCT06146231
Title: Motiva Flora® Tissue Expander as a Support for the Creation of an Autologous Adipose Matrix for Hybrid Breast Reconstruction: a Pivotal Study
Brief Title: Motiva Flora® Aesthetic Breast Recon® Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Establishment Labs (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-001000
Record Dates: First submitted 2023-11-02; First posted 2023-11-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Mammaplasty; Breast Cancer; Poland Syndrome
Keywords: Reverse expansion; Aesthetic BreastRecon™; Hybrid breast reconstruction; Implant; Autologous tissue
MeSH Terms: conditions — Breast Neoplasms; Poland Syndrome

STUDY DESIGN:
Intervention Model Description: This study is designed as a pivotal, prospective, multicentric, interventional, open-label, single-arm, non-randomized and pre-market clinical investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Motiva Flora® Tissue Expander — This hybrid breast reconstruction involves a stage in which the tissue expander (Motiva Flora®) is used as intended for a conventional expansion. After achieving the desired volume, it is deflated in a controlled way to proceed with the execution of serial fat grafting procedures (reverse expansion). This also means the expander is implanted longer than indicated on its current Directions For Use. Once the reverse expansion is complete, the expander is replaced with a long-term breast implant.
  Motiva Implants Ergonomix2® Sterile Silicone Breast Implants will be used as per Standard of Care under the CE marked indication.
  To obtain the safest, most natural, and aesthetic outcomes, Ergonomix2® breast implants have been selected as the standard silicone breast implants for this study.
  Other Names: Motiva Implants Ergonomix2® Sterile Silicone Breast Implants

SUMMARY:
The present study will be based on a hybrid breast reconstruction approach with initial skin expansion using the Motiva Flora® Tissue Expander followed by a serial fat grafting session and a final step that includes the placement of a permanent breast implant Ergonomix2®.

ELIGIBILITY:
Inclusion Criteria:

1. Genetically female, aged 18 years or older.
2. Subjects who had provided written informed consent form.
3. The participant needs tissue expansion as part of breast reconstruction treatment, which may include immediate reconstruction.
4. Clinical condition to allow reverse expansion breast reconstruction, at the investigator's discretion.
5. Sufficient fat in donor sites (abdomen, gluteus, hips, and thighs) per plastic surgeon criteria.
6. Complete radiotherapy and chemotherapy at least one year before surgery.
7. BMI between 18.5 and 30.0 (average classified weight).
8. Physical and cognitive capacity to understand and follow the surgeon's recommendations.
9. To be able and willing to comply with all study requirements, including attending follow-up appointments.

   Only Sub study participants
10. Provide additional consent to undergo an MRI with contrast.

Exclusion Criteria:

1. Current pregnancy or lactation, or full-term pregnancy or lactation at any point during the clinical investigation.
2. Abnormal hematological and biochemical values after chemotherapy.
3. High surgical risk according to the investigator.
4. Breast width larger than 18 cm
5. Tumor residues in or near the area where tissue expansion is performed.
6. Subjects with metastatic breast cancer
7. Significant Breast ptosis or poor skin quality
8. Participants who do not have adequate tissue at the intended site for expansion, at the surgeon's discretion, due to previous radiotherapy, ulceration, vascular involvement, history of impaired wound healing, or mastectomy scar deformity.
9. Inadequate chest wall tissue due to damage caused by radiotherapy, tight skin grafts, or radical resection of the pectoralis major muscle.
10. Current or previous infection in the area where the expansion occurs.
11. Any condition that impedes magnetic resonance imaging (MRI), including implanted metal device, claustrophobia, or other ailments that would prohibit MRI scan.
12. Presence of autoimmune diseases such as lupus or scleroderma, or immunocompromised participants due to immunosuppressive or steroid therapy.
13. History of silicone sensitivity.
14. Active smokers
15. Previous attempts of breast reconstruction
16. Subjects who, in the opinion of the investigator, are considered part of any vulnerable population
17. Subjects with affiliation to the Sponsor, sites or investigators, including relatives.
18. Participants who do not live in the procedure's country make it impossible to assist in follow-up visits.
19. Subjects who are participating in other investigation(s) which may affect the outcomes or ability to comply follow-up requirements of this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Total adverse envent rate | 46 months
  This variable will be assessed by the total incidence, seriousness, severity, causal relationship with the device, measure(s) taken for resolution, outcome, and duration of the various adverse events (AEs) reported during the surgery and follow-up period. The incidence of AEs, in terms of percentage, will be evaluated statistically with a 95% confidence interval. The analysis of the AEs will include:
  * All AEs reported during the time period in which Motiva Flora® TE remains implanted (up to a maximum of 16 months)
  * All AEs reported during the conduct of the whole clinical investigation (reconstruction process and 24 months follow-up)

SECONDARY OUTCOMES:
Surgeon's overall satisfaction | 46 months
  Surgeon's overall satisfaction with reconstruction process and results according to the Global Aesthetic Improvement Scale (GAIS), a 5-point Likert scale: 1) Worse (The appearance is worse than the original condition); 2) No change (The appearance is essentially the same as the original condition); 3) Improved (Obvious improvement in appearance from the initial condition, but a touch-up or retreatment is indicated); 4) Much improved (Marked improvement in appearance from the initial condition, but not completely optimal for this patient. A touch-up would slightly improve the result) and 5) Very much improved (Optimal cosmetic result for the implant in this patient).
Patient's anxiety and depression | 46 months
  Patient's anxiety and depression using the HADS (The Hospital Anxiety Depression Scale)
Patient's satisfaction and quality of life impact | 46 months
  Quality of life and satisfaction levels will be assessed using validated international tool Breast-Q.
Device's performance: Device integrity | 6-16 months
  Percentage of Tissue Expander devices found without any damage at explantation.
Changes in breast volume | 46 months
  Percentage of cases where enlargement of the initial breast volume was achieved after the fat grafting process and changes in vascularity of the filled zone documented. after the fat grafting process.
Changes in breast vascularity | 46 months
  Percentage of cases where changes in vascularity of the filled zone were documented after the fat grafting process.

CONTACTS AND LOCATIONS:
Locations (4):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Hospital Universitario San Ignacio, Bogotá, Colombia
- Hospital UNIBE, San José, Costa Rica
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No